CLINICAL TRIAL: NCT05352594
Title: The Brain Activity Changes in Persons With Low Back Pain: From Subacute to Chronic
Brief Title: The Brain Activity Changes in the Development of Chronic Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Ray-Yau Wang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: YM111017E
Record Dates: First submitted 2022-04-18; First posted 2022-04-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: Pain Chronicity; Low Back Pain; Electroencephalography; Brain Activity
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Low Back Pain: The participants whose low back pain intensity score ≥2 by numeric pain rating scale at 24-week follow-up.
- Recovered Low Back Pain: The participants whose low back pain intensity score <1 by numeric pain rating scale at 24-week follow-up.

SUMMARY:
The purpose of this longitudinal exploratory prospective study is to investigate the brain changes in the development of chronic low back pain.

DETAILED DESCRIPTION:
Background and Purpose: Chronic low back pain (cLBP) is an adverse symptom not only to individuals but also to society. It impacts negatively on multiple aspects, such as physical activities, functional ability, quality of life and psychological status. Moreover, cLBP causes economic burden to both individuals and society. However, not all low back pain progresses to chronic condition. Cross-sectional studies have shown brain activated differently in people with cLBP as compared with healthy ones during rest and movement. In addition, lower cortical excitability or stronger functional connections between medial prefrontal cortex and nucleus accumbens were observed in those becoming cLBP according to previous longitudinal studies. Also, image studies have shown a shift in brain regions from pain related areas to those that control emotion and memory. According to these results, the brain activity is related to the persistence of pain. However, how brain activity changes during the chronicity of low back pain is still not fully understood. Therefore, the purpose of present study is to compare the brain changes in people with LBP with or without pain chronicity.

Methods: This is a longitudinal exploratory prospective study. Demographic data will be collected at baseline. The outcomes will be measured at entry of the study and at 24 weeks post-pain. Outcomes include pain intensity which is rated by Numerical rating scale(NRS), and brain activities which is recorded by electroencephalography (EEG) during resting and movement conditions.

Statistical analysis: According to the NRS at 6 month post-pain, the participants whose NRS sore ≥ 2 will be grouped in the cLBP group and those NRS ≤ 1 will be grouped in the recovered low back pain (rLBP) group. Two-way ANOVA with repeated-measures and Tukey's post hoc test will be used to analyze the differences between time and between groups. The changes of pain intensity during movement will be used as confounder for the analysis. Statistical significance is set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age≧ 20 y/o
* This is the 1st episode of low back pain in the past year
* Pain in the region of the lower back (bound by the thoracolumbar junction superiorly, and by the gluteal fold inferiorly)
* Pain duration < 12 weeks
* Average pain intensity in the past 7 days is ≧ 3/10 (Numeric Rating Scale)
* Mini-Mental State Examination ≧ 24

Exclusion Criteria:

* Pain onset duration < 7 days
* History of chronic pain
* Pain area other than the specify area
* Any systematic disease, fracture or cancer
* Present any neurological sign related to pain
* Infection
* Received any brain or spine surgeries, hip arthroplasty or any other kind of surgeries in the past 3 months
* Diagnosed with any neurological or psychological disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population from community and local clinics will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity at the enrollment | at the enrollment
  The average pain intensity in the past week will be measured by numeric rating scale (NRS). NRS is a 11-point rating scale (0 represents "no pain" and 10 represents "worst pain imaginable").
Pain Intensity at 24-week follow-up | at 24-week follow-up
  The average pain intensity in the past week will be measured by numeric rating scale (NRS). NRS is a 11-point rating scale (0 represents "no pain" and 10 represents "worst pain imaginable").
Brain Activity Change from enrollment to 6-month follow-up | at the enrollment and 24-week follow-up
  Participants' brain activity will be measured by electroencephalography (EEG) during functional reaching activity to assess the brain changes.
Pain intensity during functional reaching task at the enrollment | at the enrollment
  The pain intensity during functional reaching task will be measured by numeric rating scale (NRS). NRS is a 11-point rating scale (0 represents "no pain" and 10 represents "worst pain imaginable").
Pain intensity during functional reaching task at 24-week follow-up | at 24-week follow-up
  The pain intensity during functional reaching task will be measured by numeric rating scale (NRS). NRS is a 11-point rating scale (0 represents "no pain" and 10 represents "worst pain imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No